CLINICAL TRIAL: NCT02315079
Title: Point of Care Testing of Inflammatory Markers in Tears
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201400775
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Dry Eye Syndrome
Keywords: Ocular Inflammation; Matrix Metalloproteinase 9
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — de-identified tear samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Eye inflammation: This group will have a regular eye exam with the collection of tears. In addition, a the Ocular Surface Disability Index Survey of National Eye Institute Visual Functioning Questionnaire- 25 may be administered.
  Interventions: Other: Eye inflammation
- Without eye inflammation: This group will have a regular eye exam with the collection of tears.
  Interventions: Other: Without eye inflammation

INTERVENTIONS:
Other: Eye inflammation — This group will have a regular eye exam with the collection of tears. In addition, a the Ocular Surface Disability Index Survey of National Eye Institute Visual Functioning Questionnaire- 25 may be administered.
  Groups: Eye inflammation
Other: Without eye inflammation — This group will have a regular eye exam with the collection of tears.
  Groups: Without eye inflammation

SUMMARY:
To evaluate the use of a point of care device to measure markers of inflammation in various eye conditions. In particular, matrix metalloproteinase-9 (MMP-9) will be measured. MMP-9 is an enzyme that plays a role in inflammation. The value obtained with the point of care device will be correlated with values obtained using gel electrophoresis to measure MMP-9 from the same sample. These data will be compared to clinical exam findings and questionnaires to help the investigators better understand the role of this marker of inflammation in eye diseases and possibly improve diagnostic abilities.

DETAILED DESCRIPTION:
As a participant in the study a sample of tears will be collected in a non-invasive manner by sitting comfortably at the slit lamp (a slit lamp is the standard device used to examine the eye and merely requires the participant to sit upright and place their chin on a chin rest and their forehead up against the slit lamp apparatus). The participant will then be asked to look upwards and while gently lowering the lower eyelid, a sterile blunt glass pipette will be used to collect tears from the natural tear lake (the tear lake is a reservoir of tears that sits on the surface of the eye and above the lower eyelid). Collected tears will then be taken for analysis of inflammatory markers.

In addition, a survey to evaluate the symptoms and the symptoms impact daily life (Ocular Surface Disability Index Survey of National Eye Institute Visual Functioning Questionnaire- 25).

ELIGIBILITY:
Inclusion Criteria:

* Patients that present to clinic for evaluation. Patients with and without evidence of eye inflammation will be eligible for this study.

Exclusion Criteria:

* Patients outside the age limits will not be eligible for the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-90 years of age that present to our North Central Florida Tertiary Referral University Eye Clinics for evaluation. Patients with and without evidence of eye inflammation will be eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Measurement of matrix metalloproteinase-9 in tears | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sonal Tuli, MD, Principal Investigator — University of Florida, Department of Ophthalmology
Locations (1):
- University of Florida, Department of Ophthalmology, Gainesville, Florida, United States